CLINICAL TRIAL: NCT02164747
Title: Assessment of Teleconsulting in Nursing Homes to Avoid Transportations to the Emergency Units
Acronym: TMG91
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence Regionale de Sante d'Ile de France (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLM-TMG91
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Nursing Homes Residents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control group before telemedicine: Residents of nursing homes without telemedicine before implementation of telemedicine in nursing homes with telemedicine
- Control group after telemedicine: Residents of nursing homes without telemedicine after implementation of telemedicine in nursing homes with telemedicine
- Exposed group, before telemedicine: Residents of nursing homes with telemedicine prior implementation of telemedicine
- Exposed group, after telemedicine: Residents of nursing homes with telemedicine after implementation of telemedicine
  Interventions: Device: Residents of nursing homes with telemedicine after implementation of telemedicine

INTERVENTIONS:
Device: Residents of nursing homes with telemedicine after implementation of telemedicine
  Groups: Exposed group, after telemedicine

SUMMARY:
The purpose of this study is to determine whether teleconsulting would be effective and cost-effective by reducing the patients transportations and the use of emergency units for nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* All residents of selected nursing homes

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2012-01; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Within 1 year after start of the study

SECONDARY OUTCOMES:
Patient transportation to a emergency unit | Within 1 year after start of the study
Number of hospitalizations | Within 1 year after start of the study
Global costs | Within 1 year after start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Durand-Zaleski, MD, PhD, Principal Investigator — DRCD URC Eco. Assistance Publique, Hôpitaux de Paris
Locations (5):
- France (5):
  - Résidence La Gentilhommière, Boussy-Saint-Antoine
  - Résidence Les Tisserins, Évry
  - Résidence Notre Dame d'Espérance, Milly-la-Forêt
  - Le Centenaire, Pussay
  - Résidence de l'Orge, Saint-Germain-lès-Arpajon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidholm K, Ekeland AG, Jensen LK, Rasmussen J, Pedersen CD, Bowes A, Flottorp SA, Bech M. A model for assessment of telemedicine applications: mast. Int J Technol Assess Health Care. 2012 Jan;28(1):44-51. doi: 10.1017/S0266462311000638. PMID 22617736
- [Derived] Charrier N, Zarca K, Durand-Zaleski I, Calinaud C; ARS Ile de France telemedicine group. Efficacy and cost effectiveness of telemedicine for improving access to care in the Paris region: study protocols for eight trials. BMC Health Serv Res. 2016 Feb 8;16:45. doi: 10.1186/s12913-016-1281-1. PMID 26857558